CLINICAL TRIAL: NCT02775383
Title: The National Myelodysplastic Syndromes Natural History Study
Brief Title: The National Myelodysplastic Syndromes (MDS) Study
Acronym: MDS
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NHLBI-MDS
Record Dates: First submitted 2016-05-02; First posted 2016-05-17 (Estimated); Last update posted 2026-02-03 (Actual); Status verified 2025-11

CONDITIONS: Myelodysplastic Syndromes (MDS)
Keywords: National MDS Study; MDS; Idiopathic; cytopenia; cytopenias; ICUS; MDS/MPN; Myeloproliferative Neoplasm; Biorepository
MeSH Terms: conditions — Myelodysplastic Syndromes; Cytopenia; Myeloproliferative Disorders | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Years
Biospecimen Retention: Samples With DNA — bone marrow, peripheral blood, serum, plasma, eyebrow hairs with attached follicles, buccal cells, skin biopsy
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Longitudinal: Participants with MDS, MDS/MPN overlap disorder, AML <30% blasts without core binding factor or acute promyelocytic leukemia, ICUS, or at risk based on select karyotypic or genetic abnormalities
  Interventions: Other: Therapeutic
- Cross-sectional: Participants who do not have MDS, MDS/MPN overlap disorder, or ICUS and have the baseline visit only
  Interventions: Other: Therapeutic

INTERVENTIONS:
Other: Therapeutic — Observational Study

SUMMARY:
Multi-center study enrolling patients suspected or newly diagnosed with myelodysplastic syndromes (MDS), myelodysplastic syndromes/myeloproliferative neoplasms (MDS/MPN) overlap disorder, or idiopathic cytopenia of undetermined significance (ICUS). Participants will be followed long term. Clinical data, blood, and tissue samples will be collected to establish a biorepository to facilitate the study of the natural history of MDS.

DETAILED DESCRIPTION:
Multi-center, prospective cohort study enrolling patients from centers in the National Cancer Institute (NCI) National Clinical Trials Network (NCTN) and NCI Community Oncology Research Program (NCORP). The accrual period is 5+ years. After central pathology review of registered participants, approximately 2,000 cases of MDS or MDS/MPN overlap disorders, and 500 cases of ICUS will be identified for the longitudinal study cohort and up to 1000 cases will be identified for the cross-sectional cohort. No more than 3500 total participants will be registered. Participants in the longitudinal cohort may be followed for life.

The goal of the National MDS Study is to establish a publicly available resource to facilitate the study of MDS natural history. This will be accomplished through: 1) Creation of a multi-institutional, longitudinal collection of consistently processed and clinically well-annotated blood and tissue specimens collected prospectively from participants with MDS and participants with idiopathic cytopenia of undetermined significance (ICUS); and 2) Support for investigator-initiated studies of MDS that will have high-impact for MDS patients, including basic science, clinical, health outcomes and epidemiological research.

ELIGIBILITY:
Inclusion Criteria:

* Suspected (e.g., persistent unexplained cytopenia, circulating peripheral blasts etc.) MDS or MDS/MPN overlap disorders and undergoing diagnostic work-up with planned bone marrow assessments, or diagnosed with de novo or therapy-related MDS within 12 months of enrollment per the World Health Organization (WHO) criteria1 and undergoing clinical evaluation and planned bone marrow assessments to confirm MDS or to evaluate disease status
* Bone marrow aspirate expected to be performed within 1 week of registration, and in all cases must be performed no later than 4 weeks after enrollment
* Age 18 or older
* If anemic without prior MDS diagnosis, B12 level, serum folate, mean corpuscular volume (MCV), red cell distribution width (RDW), ferritin, and iron studies (Iron, total iron-binding capacity (TIBC) test, and percent saturation) must be performed within prior 6 months.

Exclusion Criteria:

* Prior treatment for MDS at entry and through the time of the entry bone marrow aspirate
* Treatment with hematopoietic growth factors in prior 6 months
* Diagnosis of a solid tumor or hematologic malignancy within two years prior to enrollment except for in situ cancer of the skin (basal or squamous cell), cervix, bladder, breast, or prostate
* Treatment with radiation therapy in the two years prior to registration
* Non-hormonal treatment for malignancy within the two years prior to registration
* Established hereditary bone marrow failure syndrome
* Known primary diagnosis of aplastic anemia, classical paroxysmal nocturnal hemoglobinuria, amegakaryocytic thrombocytopenic purpura, or large granular lymphocyte leukemia
* Enrolled in the Connect® MDS/AML Disease Registry (NCT01688011)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected MDS or MDS/MPN overlap disorder who are undergoing diagnostic workup and bone marrow assessments, and patients diagnosed with MDS within 6-months of enrollment and undergoing clinical evaluation and bone marrow assessments to confirm MDS or evaluate disease status
Sampling Method: Non-Probability Sample
Enrollment: 2115 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients dying | Through study completion, an average of 3 years
  Deaths will be reported on study case report forms

SECONDARY OUTCOMES:
Number of participants progressing to Acute Myeloid Leukemia (AML) | Through study completion, an average of 3 years
  Progression to AML will be reported on study case report forms

CONTACTS AND LOCATIONS:
Overall Officials: Mikkael Sekeres, MD, MS, Study Chair — University of Miami; Amy DeZern, MD, MHS, Study Chair — Johns Hopkins University
Locations (281):
- United States (280):
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente - South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Tibor Rubin VA Medical Center, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente-Cadillac, Los Angeles, California
  - Va Palo Alto Health Care System, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Veterans Affairs Connecticut Healthcare System-West Haven Campus, West Haven, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Indian River Medical Center, Vero Beach, Florida
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Northside Hospital - Duluth, Duluth, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Suburban Hematology Oncology Associates - Snellville, Snellville, Georgia
  - Queen's Cancer Center - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - OnCare Hawaii - Liliha, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Cancer Care Specialists of Central Illinois - Decatur, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - AMITA Health Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - AMITA Health Cancer Institute and Outpatient Center, Hinsdale, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Specialists of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare - Peoria, Peoria, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Cancer Center of Kansas - Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas - Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Waldo County General Hospital, Belfast, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Biddeford, Biddeford, Maine
  - Stephens Memorial Hospital, Norway, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Sanford, Sanford, Maine
  - Maine Medical Partners-South Portland, South Portland, Maine
  - York Hospital, York Village, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Ascension Providence Hospitals - Southfield, Southfield, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic - Rolla - Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare-Sletten Cancer Institute, Great Falls, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Oakey, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Mountainview, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Veterans Administration New Jersey Health Care System, East Orange, New Jersey
  - Inspira Medical Center Woodbury, Woodbury, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Glens Falls Hospital, Glens Falls, New York
  - North Shore University Hospital, Lake Success, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Phelps Memorial Hospital Center, Sleepy Hollow, New York
  - Montefiore Medical Center - Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - James J Peters VA Medical Center, The Bronx, New York
  - Mission Hospital, Asheville, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Fairview, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Kaiser Permanente Northwest, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital-Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Easton Hospital, Easton, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Geisinger Medical Center - Cancer Center Hazleton, Hazleton, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology - Lewisburg, Lewisburg, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Phoenixville Hospital, Phoenixville, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - Geisinger Cancer Services - Pottsville, Pottsville, Pennsylvania
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Ralph H Johnson VA Medical Center, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health System Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health System Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health System Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health System Cancer Institute - Butternut, Reidville, South Carolina
  - Prisma Health System Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Prisma Health System Cancer Institute - Spartanburg, Spartanburg, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Monument Health Rapid City Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Augusta Health Center for Cancer and Blood Disorders, Fishersville, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Ascension Southeast Wisconsin Hospital-Elmbrook Campus, Brookfield, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Medical Center - EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fontana, Wisconsin
  - Ascension Saint Francis-Reiman Cancer Center, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - William S Middleton VA Medical Center, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Vince Lombardi Cancer Clinic-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center - Marshfield, Marshfield, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center - Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Ascension Medical Group Southeast Wisconsin-Mayfair Road, Wauwatosa, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Clinic-Weston Center, Weston, Wisconsin
- Shaare Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Derived] Abel GA, Hebert D, Lee C, Rollison D, Gillis N, Komrokji R, Foran JM, Liu JJ, Al Baghdadi T, Deeg J, Gore S, Saber W, Wilson S, Otterstatter M, Thompson J, Borchert C, Padron E, DeZern A, Cella D, Sekeres MA. Health-related quality of life and vulnerability among people with myelodysplastic syndromes: a US national study. Blood Adv. 2023 Jul 25;7(14):3506-3515. doi: 10.1182/bloodadvances.2022009000. PMID 37146263
- [Derived] DeZern AE, Goll JB, Lindsley RC, Bejar R, Wilson SH, Hebert D, Deeg J, Zhang L, Gore S, Al Baghdadi T, Maciejewski J, Liu J, Padron E, Komrojki R, Saber W, Abel G, Kroft SH, Harrington A, Grimes T, Reed H, Fulton RS, DiFronzo NL, Gillis N, Sekeres MA, Walter MJ. Utility of targeted gene sequencing to differentiate myeloid malignancies from other cytopenic conditions. Blood Adv. 2023 Jul 25;7(14):3749-3759. doi: 10.1182/bloodadvances.2022008578. PMID 36947201
- See also: Website for The National Myelodysplastic Syndromes Natural History Study — http://thenationalmdsstudy.net/